CLINICAL TRIAL: NCT00948519
Title: Laser Microbial Killing With Photo Activated Agents
Brief Title: Laser Assisted Treatment of Chronic Sinusitis With and Without Light Activated Agents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York Head & Neck Institute (Other)
Collaborators: Valam Corp. (Industry)
Responsible Party: Yosef Krespi, Victor Kizhner, St.Luke's-Roosevelt
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SLR 09-005
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2009-07

CONDITIONS: Rhinosinusitis
Keywords: Rhinosinusitis, sinusitis, chronic, nasal polyps, phototherapy, laser,laser therapy, antibiotic, safety laser, ICG, indocyanine green; Chronic Rhinosinusitis with or without nasal polyposis
MeSH Terms: conditions — Rhinosinusitis; Sinusitis; Bronchiolitis Obliterans Syndrome; Nasal Polyps | interventions — Lasers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser + ICG (Experimental): ICG arm- will be defined as local application on a pledget soaked with ICG with a concentration of 200µg, upon removal of the pledget a NIR diode laser set at 6W with light emittance introduced intranasally with a 30mm diffuser fiber capable of radiating light circumferentially allowing the light energy to reach all treatable areas. Laser will be activated for 180 seconds. Assuming an approximate radius of the nasal cavity is 3mm, energy density will be around 200J/cm². Treatment will be repeated twice, 5-7 day apart. Cultures will be collected at the end of all treatments
  Interventions: Device: Laser + ICG
- Laser only (Active Comparator): same as above, without ICG
  Interventions: Device: Laser only

INTERVENTIONS:
Device: Laser + ICG — ICG arm- will be defined as local application on a pledget soaked with ICG with a concentration of 200µg, upon removal of the pledget a NIR diode laser set at 6W with light emittance introduced intranasally with a 30mm diffuser fiber capable of radiating light circumferentially allowing the light energy to reach all treatable areas. Laser will be activated for 180 seconds. Assuming an approximate radius of the nasal cavity is 3mm, energy density will be around 200J/cm². Treatment will be repeated twice, 5-7 day apart. Cultures will be collected at the end of all treatments
  Arms: Laser + ICG
Device: Laser only — same only without ICG
  Arms: Laser only

SUMMARY:
Chronic rhinosinusitis (CRS) is common disorder which affects up to 13% of the US population. CRS affects numerous Quality of Life (QOL) factors including smell, sleep and communication. The common treatment for medically noncompliant CRS is Functional Endoscopic Sinus Surgery (FESS).

As the disease course is generally idle, prolonged medical treatment guidelines are for antibiotic treatment, prescribed accordingly following appropriately obtained nasal cultures, lasting weeks with or without additional topical or oral steroid treatment. While FESS success rate is a general notion, a failure rate of primary FESS is as high as 2-24%2, with a Cochrane review even suggesting that FESS though a safe procedure is of no benefit more than medical management.

With that in mind as we address the failed FESS, new bacteria emerge. The new bacteria in CRS are Coagulase-negative staphylococci were the most common isolates (36%), followed by Staphylococcus aureus (25%), Streptococcus viridans (8.3%), Corynebacterium (4.6%), and anaerobes (6.4%).

Patients not relieved by primary FESS demonstrate a significant rise in Pseudomonas and MRSA bacteria positive cultures. Moreover surgical success for patients with Staphylococcus aureus and Pseudomonas aeruginosa positive cultures is usually reduced.

Bacterial killing, by usage of light-activated agents such as Indocyanine Green (ICG) with exposure to the specific wavelength, eventually produces bacterial killing. Mechanisms primarily involved are production of reactive oxygen species (i.e. singlet oxygen and free radicals) which can then kill bacteria. ICG by itself does not have any bacterial killing effect.

Low level laser therapy (LLLT) was shown to be effective as a bactericidal by single and multiple wave exposures.

The study purpose is to treat CRS with an alternative to antibiotics, thus sparing volunteers from prolonged antibiotics use and its possible side effects, not to mention the cost and growth of resistant bacteria. We believe that by combining ICG with light or even by light alone we can produce you a beneficial effect. Although this has been shown to kill bacteria in lab or animal studies it is still investigational for humans. The study will have two arms: ICG + laser and laser only arm. ICG will be applied locally in the nasal passage (internally) followed by laser activation with a power setting of 6W. The laser will be activated with a diffuser mode meaning light of a specific known wavelength will be delivered evenly in the nasal cavity and not as a beam. Laser only treatment plan will be the same only without ICG. Volunteers will be assigned to one of the groups randomly meaning you have a 50% chance of enrolling to each treatment group. Volunteers will not know to which group. Weekly visits with a total of three visits will follow. With each visit Volunteers will receive additional treatment as the initial treatment was and a nasal culture will be taken. Volunteers will have to fill a questionnaire with each visit.

DETAILED DESCRIPTION:
A prospective randomized trial that will be performed over the period of 1 year or until 20 patients in each arm meeting inclusion criteria will be recruited. One arm will be treated with a NIR laser (ARC Lasers Gmbh, Germany) alone and another arm will have an ICG+ NIR laser treatment.

FDA approved NIR lasers in the range of 810- 980nm. FDA approved ICG (Akorn, Buffalo Grove, IL) applied locally total application will not exceed 2.5 mg Randomization method: first five volunteers will start the ICG+ laser followed by five from only laser treatment group. This will be followed by allocating one volunteer to each study arm alternatively.

Data to be collected: demographical data including age and gender, approximate duration of symptoms, culture results, SNOT 20 (QOL questionnaire) score.

Urine test will be done to rule out pregnancy prior to study enrollment. Treatment: ICG arm- will be defined as local application on a pledget soaked with ICG with a concentration of 200µg, upon removal of the pledget a NIR diode laser set at 6W with light emittance introduced intranasally with a 30mm diffuser fiber capable of radiating light circumferentially allowing the light energy to reach all treatable areas. Laser will be activated for 180 seconds. Assuming an approximate radius of the nasal cavity is 3mm, energy density will be around 200J/cm². Treatment will be repeated twice, 5-7 day apart. Cultures will be collected at the end of all treatments.

Non-ICG arm: same as above but without ICG appliance. Follow up will consist of an office visit upon end of treatment with an additional visit scheduled two weeks later Protective equipment: specifically designed eye goggles, draping preventing clothes stains from the dye

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18
* Patients with an established nasal culture of either

  * Staph aureus,
  * Strep species,
  * Pseudo monasaureginosa,
  * Proteus.mirabilis,
  * H. influenza
  * or other intranasal pathogens.

Exclusion Criteria:

* Patients without CRS,
* Patients known to have Iodide allergy or ICG allergy
* Patients scheduled for a thyroid scan
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Quality of Life improvement with disease control. Disease control without antibiotics or steroids. | 1-2 months

SECONDARY OUTCOMES:
Laser safety without compromising disease progress | immediate and late

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - St.Luke's-Roosevelt, New York Head Neck Institute, New York, New York
  - Head Neck Surgical Group, New York, New York
  - New York Head Neck Institute, New York, New York

REFERENCES:
- [Background] Omar GS, Wilson M, Nair SP. Lethal photosensitization of wound-associated microbes using indocyanine green and near-infrared light. BMC Microbiol. 2008 Jul 1;8:111. doi: 10.1186/1471-2180-8-111. PMID 18593460
- [Background] Guffey JS, Wilborn J. Effects of combined 405-nm and 880-nm light on Staphylococcus aureus and Pseudomonas aeruginosa in vitro. Photomed Laser Surg. 2006 Dec;24(6):680-3. doi: 10.1089/pho.2006.24.680. PMID 17199465